CLINICAL TRIAL: NCT05335759
Title: Coaching Programme to Improve Nurses' Perceptions of Preceptorship of Undergraduate Students: An Exploratory Trial
Brief Title: Coaching Programme for Preceptorship of Undergraduate Nurses' Students
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: CPMS
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-04

CONDITIONS: Education; Nursing
Keywords: Coaching; Preceptorship; Intervention; Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Coaching programme for improvement and development of teaching skills in preceptorship — Training program An intervention based on coaching. The strategies of this program consisted of three 6-hour sessions using case studies and role-playing for motivation towards the development of the teaching role in the preceptorship of undergraduate nursing students and debriefing and a 4-hour booster session seven months later.

SUMMARY:
Background: During the curricular practices of the Bachelor's Degree in Nursing, students are prepared to carry out an adequate transition process to the professional role. The success of this preparation depends, to a large extent, on preceptorship. In this sense, it is important that practice tutors are motivated and feel competent to teach in the clinical setting. Despite this, no studies have been found that implement and evaluate an intervention to improve nurses' perceptions of preceptorship of undergraduate nursing students.

Purpose: To evaluate the preliminary efficacy of a coaching programme to improve nurses' perceptions of preceptorship of undergraduate nursing students. Specifically, the aim is to determine the impact of the programme on nurses' perceived involvement, motivation, satisfaction, barriers and commitment to clinical mentoring.

Method: An exploratory pre-post quasi-experimental pilot study. Fifteen nurses, the total population of nurses working in the medical-surgical ward, with at least 1 year of experience in the preceptorship of students, will be recruited in June 2022. All the nurses will receive an intervention based on coaching. The strategies of this program consisted of five 6-hour sessions using case studies and role-playing simulations to work on their motivation to develop their teaching role in the preceptorship of undergraduate nursing students and debriefing and a 4-hour booster session seven months later. The IMSOC (involvement, motivation, satisfaction, obstacles and commitment) instrument was used to assess outcomes. The primary outcome was the difference in the median of nurses' involvement, motivation, satisfaction, barriers and commitment in preceptorship students pre and post-intervention (between T0-T1 and T0-T2). Changes within nurses were analyzed using the Wilcoxon test for related samples.

DETAILED DESCRIPTION:
Data collection:

Data collection was divided into three times: T0, T1 and T2. T0 corresponds to preintervention data and T1 and T2 to post-intervention data (T1 after the training and T2 after the whole intervention implementation).

IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) questionnaire. This questionnaire measures the involvement, motivation, satisfaction, obstacles and commitment of nurses in tutoring students. It is a validated instrument that shows adequate psychometric properties (overall Intraclass Correlation Coefficient (ICC) of 0.852 and internal consistency - Cronbach's α of 0.837). It consists of 33 items measured on a 5-point Likert scale (1=strongly disagree - 5=strongly agree).

Ethical considerations:

This study conformed to the principles set out in the Declaration of Helsinki and was approved by the centre's board and by the Research Ethics Committee (code 2022.044). Data custody complied with Organic Law 3/2018 on data protection (LOPDE). Informed consents were given to all participants. They were informed verbally and in writing about their free participation, the confidentiality of the data and its use for scientific purposes.

ELIGIBILITY:
* Inclusion Criteria:

  * Nurses working in the medical-surgical ward.
  * Nurses with at least one year's experience in the preceptorship of students.
  * Nurses who have voluntarily agreed to participate in the study.
* Exclusion Criteria:

  * Nurses who are not working during the time of the study (sick leave or maternity leave).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical nurses working in the medical-surgical ward during the time of the intervention evaluation were the target population from which the sample was taken.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) Questionnaire | T0 (2022 September-October)
  Nurses' involvement, motivation, satisfaction, barriers and commitment in preceptorship students
  Measurement tool: IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) Questionnaire.
  * Involvement: 8 items measured on a 5-point Likert scale [8=unsuitable - 40=excellent].
  * Motivation: 8 items measured on a 5-point Likert scale [8=unsuitable - 40=excellent].
  * Satisfaction: 6 items measured on a 5-point Likert scale [6=unsuitable - 30=excellent].
  * Obstacles: 6 items measured on a 5-point Likert scale [6=unsuitable - 30=excellent].
  * Commitment: 5 items measured on a 5-point Likert scale [5=unsuitable - 25=excellent].
IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) Questionnaire | T1 (2022 November)
  Nurses' involvement, motivation, satisfaction, barriers and commitment in preceptorship students
  Measurement tool: IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) Questionnaire.
  * Involvement: 8 items measured on a 5-point Likert scale [8=unsuitable - 40=excellent].
  * Motivation: 8 items measured on a 5-point Likert scale [8=unsuitable - 40=excellent].
  * Satisfaction: 6 items measured on a 5-point Likert scale [6=unsuitable - 30=excellent].
  * Obstacles: 6 items measured on a 5-point Likert scale [6=unsuitable - 30=excellent].
  * Commitment: 5 items measured on a 5-point Likert scale [5=unsuitable - 25=excellent].
IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) Questionnaire | T2 (2023 May)
  Nurses' involvement, motivation, satisfaction, barriers and commitment in preceptorship students
  Measurement tool: IMSOC (Involvement, Motivation, Satisfaction, Obstacles and Commitment) Questionnaire.
  * Involvement: 8 items measured on a 5-point Likert scale [8=unsuitable - 40=excellent].
  * Motivation: 8 items measured on a 5-point Likert scale [8=unsuitable - 40=excellent].
  * Satisfaction: 6 items measured on a 5-point Likert scale [6=unsuitable - 30=excellent].
  * Obstacles: 6 items measured on a 5-point Likert scale [6=unsuitable - 30=excellent].
  * Commitment: 5 items measured on a 5-point Likert scale [5=unsuitable - 25=excellent].

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Vázquez-Calatayud, PhD, Principal Investigator — University of Navarra
Locations (2):
- Spain (2):
  - Navarre, Pamplona
  - University of Navarra, Pamplona